CLINICAL TRIAL: NCT03678740
Title: Diagnostic Odyssey Survey 2
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: Columbia University (Other); United Mitochondrial Disease Foundation (Unknown); George Washington University (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NAMDC 7419
Record Dates: First submitted 2018-09-18; First posted 2018-09-20 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-03

CONDITIONS: Mitochondrial Diseases
MeSH Terms: conditions — Mitochondrial Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Odyssey 2 Survey — Odyssey2 will retain the strengths (simplicity, brevity, confidentiality, and data quality assurance measures) which made Odyssey1 successful. While Odyssey2 adds some refinements based on experience learned from Odyssey1, the basic questions are changed as little as possible to maximize comparability, and the additions are limited. Odyssey1 consisted of between 16 and 23 questions, depending on skip patterns, and took an estimated 15 minutes to complete. Odyssey2 consists of between 23 and 33 questions, depending on skip patterns and we estimate that it will take approximately 20 minutes to complete.

SUMMARY:
A previous NAMDC survey study (NAMDC 7414 - Diagnostic Odyssey Survey, referred to hereafter as Odyssey1), provided a benchmark account of the substantial challenges faced by patients in achieving a diagnosis of mitochondrial disease, and of the impact such a diagnosis has on them (Grier et al. 2018).1 This study was conducted from October 2015 through January 2016. We propose a new survey study (Odyssey2) which will provide an update, additional data collection (duration of the diagnostic odyssey), and allow assessment of next-generation DNA sequencing techniques since Odyssey1 concluded.

Odyssey2 will retain the strengths (simplicity, brevity, confidentiality, and data quality assurance measures) which made Odyssey1 successful. While Odyssey2 adds some refinements based on experience learned from Odyssey1, the basic questions are changed as little as possible to maximize comparability, and the additions are limited. Odyssey1 consisted of between 16 and 23 questions, depending on skip patterns, and took an estimated 15 minutes to complete. Odyssey2 consists of between 23 and 33 questions, depending on skip patterns and we estimate that it will take approximately 20 minutes to complete. As in Odyssey1, only patients who report, directly or through a guardian, that they have been informed by a doctor that they have a confirmed mitochondrial disorder will be eligible for Odyssey2.

DETAILED DESCRIPTION:
To gain an understanding of the "Diagnostic Odyssey" patients with mitochondrial disease undergo the Odyssey2 survey will address the following 7 questions. The first 6 are the same as in Odyssey1.

1. How much time typically elapses between when patients initially notice symptoms of a mitochondrial disorder and when they receive the diagnosis of mitochondrial disease?
2. How many physicians do patients typically see before they receive the diagnosis of mitochondrial disease?
3. What testing do patients typically undergo?
4. What other diagnoses, if any, do patients typically receive?
5. How did receiving a mitochondrial disease diagnosis impact the patient's life?
6. If the patient were to learn that their mitochondrial disease diagnosis was incorrect, what impact would that have?
7. Have any of the above changed since Odyssey1 in the RDCRN results?

Upon collection, the survey data will be stored by the Rare Diseases Clinical Research Network (RDCRN) Data Management and Coordinating Center (DMCC) at the University of South Florida.

Upon conclusion of the study period, the data will be de-identified prior to being sent to Dr. Seamus Thompson at the NAMDC Data Coordinating Center (DCC). The data will be analyzed by a team which will include Drs. Thompson, Hirano, Karaa, and Yeske; and Ms. Shepard, the project statistician. All data collected will be sent to a Federal data repository to be stored indefinitely per the current RDCRN data sharing policy.

ELIGIBILITY:
Inclusion Criteria:

-Individuals who report receiving a diagnosis of mitochondrial disease from a doctor, who are enrolled in the Rare Diseases Clinical Research Network (RDCRN) NAMDC Contact Registry

OR

-Individuals who report receiving a diagnosis of mitochondrial disease from a doctor, who are enrolled in the United Mitochondrial Disease Foundation (UMDF) Mitochondrial Disease Community Registry (MDCR)

AND

-Individuals who are able to provide consent

AND

-Individuals who are able to complete the survey

Exclusion Criteria:

-Individuals who do not report receiving a diagnosis of mitochondrial disease from a doctor, who are enrolled in the Rare Diseases Clinical Research Network (RDCRN) NAMDC Contact Registry.

OR

-Individuals who do not report receiving a diagnosis of mitochondrial disease from a doctor, who are enrolled in the United Mitochondrial Disease Foundation (UMDF) Mitochondrial Disease Community Registry (MDCR).

OR

-Individuals who are unable to provide consent

OR

-Individuals who are unable to complete the survey

Max Age: 99 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Individuals will be recruited from the RDCRN NAMDC Contact Registry or UMDF Mitochondrial Disease Community Registry (MDCR) who report that they have been informed by a doctor that they have a confirmed mitochondrial disorder.
Sampling Method: Non-Probability Sample
Enrollment: 336 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
Duration of the Diagnostic Odyssey | 4 months
  The primary outcome measure is to provide an update, perform additional data collection (duration of the diagnostic odyssey), and allow assessment of next-generation DNA sequencing techniques since Odyssey1 concluded.

CONTACTS AND LOCATIONS:
Overall Officials: John Thompson, PhD, Study Chair — Columbia University
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No